CLINICAL TRIAL: NCT06717724
Title: Complementary Treatment With Procaine Periarticular Injections for Pain Reduction and Functional Improvement in Elderly Individuals With Osteoarthritis
Brief Title: § Procaine Periarticular Injections for Pain Reduction in Elderly With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sf Luca Chronic Disease Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SfLucaCDHProcaine
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-02

CONDITIONS: HIP AND KNEE OSTEOARTHRITIS; Geriatric Assessment; Geriatric Depression
Keywords: procaine; infiltration; geriatric assessment; periarticular injections; gerovital h3; geriatric depression; hip osteoarthritis; knee osteoarthritis; ana aslan; physical therapy; activities of daily living (ADL); instrumental activities of daily living (IADL)
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants are divided into an experimental group that receives the basic treatment combined with the intervention and one control group that receives the basic treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants in the experimental arm received daily periarticular injections of procaine complex solution (5 ml containing 100 mg procaine hydrochloride) over a 10-day period. All injections were administered using sterile technique. Prior to treatment, sensitivity to procaine hydrochloride was assessed with a subcutaneous test dose (0.5 ml)
  Interventions: Drug: Periarticular Procaine Injection (PAPI); Other: Kinesiotherapy
- Control (Active Comparator): Participants received only physical therapy without procaine injections.
  Interventions: Other: Kinesiotherapy

INTERVENTIONS:
Drug: Periarticular Procaine Injection (PAPI) — Participants will receive periarticular 5 ml procaine injections targeting painful joints for 10 consecutive days alternating between knee- and/or hip joints
  Arms: Experimental
Other: Kinesiotherapy — Kinesiotherapy

SUMMARY:
§ The goal of this clinical trial is to assess the effect of periarticular procaine injections combined with physical therapy on joint pain in individuals 65 and older suffering from osteoarthritis of the hip or the knee. The main question it aims to answer is: Is procaine effective in decreasing joint pain?

Researchers will compare procaine injections combined with physical therapy to physical therapy only to evaluate whether or not procaine helps decrease joint pain.

Participants will:

Undergo procaine periarticular injections and physical therapy Assess their symptoms and pain using scales and tests provided

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the safety and efficacy of procaine complex injections in managing pain and improving functional capacity in elderly patients with osteoarthritis in the knee and/or hip. The study enrolled 178 patients aged 65 and older, who were randomly assigned to receive either physical therapy combined with periarticular procaine injections or physical therapy alone. Pain levels were assessed using the Visual Analogue Scale (VAS), and functional capacity was evaluated using the Lequesne Index, Activities of Daily Living (ADL), Instrumental Activities of Daily Living (IADL), and other geriatric assessment tools. Results indicated significant pain reduction and functional improvement in the procaine group, highlighting a safe alternative treatment to surgery for older adults with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 and older diagnosed with knee or hip osteoarthritis per the American College of Rheumatology criteria. Must exhibit radiographic evidence of OA and experience persistent joint pain

Exclusion Criteria:

* Individuals with Alzheimer's, severe depression, cancer, or other severe health conditions, and those with allergies to procaine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 203 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Pain Levels | Baseline to Day 10
  Change in Pain Level on Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Functional Improvement | Baseline to Day 10
  Change in Lequesne Index Score
ADL and IADL Scores | Baseline to Day 10
  Changes in Activities of Daily Living and Instrumental ADL scores
Geriatric Depression Scale | Baseline to Day 10
  Change in Depression Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sorina Maria Aurelian, Principal Investigator — "Carol Davila" University of Medicine and Pharmacy Geriatrics and Gerontology Clinic, "Sf. Luca" Chronic Disease Hospital Bucharest
Locations (1):
- "Sf. Luca" Chronic Disease Hospital, Bucharest, Romania